CLINICAL TRIAL: NCT01586338
Title: A Multicenter, Prospective, Open-label, Single Arm Study of the Efficacy and Safety of Synvisc® (Hylan G-F 20) in Chinese Subjects With Symptomatic Osteoarthritis of the Knee(s)
Brief Title: A Study of the Efficacy and Safety of Synvisc® in Chinese Subjects With Symptomatic Osteoarthritis of the Knee(s)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNVIL06244; U1111-1129-3321 (Other: UTN); EFC13912 (Other: Sanofi)
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — hylan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synvisc (Experimental): Three intra-articular (IA) injections of Synvisc (2.25 ml glass syringe containing 16 mg hylan G-F 20) at intervals of one week. The total duration of observation was 26 weeks.
  Interventions: Drug: Hylan G-F 20

INTERVENTIONS:
Drug: Hylan G-F 20 — Intra-articular injection (pre-filled glass syringe)
  Other Names: Synvisc®

SUMMARY:
Primary Objective:

* To evaluate the change of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 subscore (walking pain) at 26 weeks compared to the Baseline score
* To evaluate the safety using the incidence, severity, seriousness, relatedness, and frequency of all treatment emergent Adverse Events (AEs)

Secondary Objectives:

* To evaluate the change in WOMAC A1 subscore (walking pain) between baseline and weeks 8, and 12
* To evaluate the change in WOMAC A, B and C score between baseline and weeks 8, 12 and 26
* To evaluate the change in Patient Global Assessment (PTGA) score between baseline and weeks 8, 12 and 26
* To evaluate the change in Clinical Observer Global Assessment (COGA) score between baseline and weeks 8, 12 and 26
* To evaluate the change in concomitant Osteoarthritis (OA) therapy over 26 weeks and between baseline and weeks 1, 2, 8, 12 and 26

DETAILED DESCRIPTION:
Duration of study period for each participants was 26-28 weeks.

ELIGIBILITY:
Inclusion criteria :

1. The participants had a diagnosis of OA of the Target Knee confirmed by recent X-Ray (mild to moderate joint space narrowing and/or osteophytes predominant in the tibiofemoral compartment)
2. WOMAC A1 baseline 100 mm Visual Analog Score (VAS) between 40-80 mm (moderate or severe walking pain) in the Target knee
3. Participants with bilateral disease included in the study with the below strict conditions:

   * Only one knee included in the efficacy assessment and considered the Target Knee (The worst knee by the WOMAC A1 pain scale should be selected). The selected knee must meet the inclusion and exclusion criteria
   * The non-target knee might also be treated with Synvisc® and did not need to meet the Kellgren-Lawrence (KL) grade knee specific inclusion criteria described above. The other criteria applied, and included in safety assessment
4. Pre-menopausal female participants had a negative urine pregnancy test and continue to use a medically acceptable form of contraception for the duration of the study. Otherwise, females had been surgically sterile, or postmenopausal (as documented in medical history) for at least 1 year

Exclusion criteria:

1. Significant (requiring surgical correction) valgus or varus deformity of the knee, ligamentous laxity, or meniscal instability
2. Concomitant inflammatory or any other disease/condition which might affect joints (e.g., rheumatoid arthritis, metabolic bone disease, psoriasis, gout, pseudogout, chondrocalcinosis etc)
3. History of sepsis in any joint or any clinical concern for a sub-acute infectious process in the target joint
4. History of surgery in the target knee (if done < 6 months)
5. Planned surgery on any lower extremity joint
6. Presence of clinically significant venous or lymphatic stasis in the leg(s)
7. Clinically apparent tense effusion or inflammation at the target knee
8. Skin disease or infection in the area of the injection site
9. Any musculoskeletal condition that would impede measurement of efficacy at the target knee
10. Pregnant or lactating women
11. Hypersensitivities to avian proteins and/or any components of hyaluronan-based injection
12. Treatment with any Hyaluronic Acid (HA) or derivatives in the previous 6 months.
13. Treatment with Intra-Articular (IA) steroid in the previous 3 months
14. Any contra-indication to IA injection e.g., anticoagulant therapy or clinical concern for potential coagulopathy (e.g. liver disease)
15. Any significant medical condition (e.g., significant psychiatric or neurological disorders, active alcohol/drug abuse, etc), any medical condition that is unstable/poorly controlled or other factor (e.g., planned relocation) that the Investigator felt would interfere with study evaluations and study participation

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 centers in China. A total of 237 participants were enrolled between March 09, 2012 and February 28, 2013.
Pre-assignment Details: Of 237 enrolled participants 232 participants were treated. 5 participants were excluded from total enrolled (3 participant due to informed consent filled by family, and 2 participant due to no efficacy data after treatment).
Period: Overall Study
Arm/Group | Synvisc
Started | 237
Completed | 229
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by participant | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- Synvisc: Three IA injections of Synvisc (2.25 ml glass syringe containing 16 mg hylan G-F 20) at intervals of one week. The total duration of observation was 26 weeks.
Arm/Group | Synvisc
Number analyzed (Participants) | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 Subscore (Walking Pain) at Week 26
Description: WOMAC is health status measure questionnaire of twenty-four questions comprising 3 subscales (pain, stiffness and physical function). WOMAC A1 (walking pain) was measured on a scale of 0-100 mm, where lower score represents lower pain and higher score represents higher pain.
Time Frame: Baseline, Week 26 (missing data imputed by Last Observation Carried Forward [LOCF])
Population: Full Analysis Set (FAS) included all participants who received at least one injection of Synvisc®. 5 participants were excluded from total enrolled (3 participant due to informed consent filled by family, and 2 participant due to no efficacy data after treatment).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Synvisc
Number analyzed (Participants) | 232
mm | -33.0 (17.71)
Statistical Analysis 1: Comparison: Synvisc; Test type: Superiority or Other; p < 0.0001, Paired t-test — Threshold for significance = 0.05
Statistical Analysis 2: Comparison: Synvisc; Test type: Superiority or Other; p < 0.0001, Sign Rank Test

2. Primary Outcome: Overview of Adverse Events (AE)
Description: An AE could be any unfavorable and unintended symptom, sign, disease or condition, or test abnormality whether or not considered related to the investigational product. A serious adverse event (SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs (TEAE): AEs that developed/worsened during the 'on treatment period' (from first dose of study drug until the end of study period). Category "AE" included participant with both serious and non-serious AE.
Time Frame: Up to Week 26
Population: Safety Set included all participants who received at least one injection of Synvisc.
Measure: Number; unit: percentage of participants
Arm/Group | Synvisc
Number analyzed (Participants) | 237
percentage of participants
  AEs | 27.8
  Treatment-emergent AEs | 27.8
  Treatment-emergent SAEs | 1.7
  Treatment-emergent AEs Lead to Discontinuation | 0.4

3. Secondary Outcome: Change From Baseline in WOMAC A1 Subscore (Walking Pain) at Week 8 and 12
Description: as for outcome 1
Time Frame: Baseline, Week 8 and Week 12 (missing data imputed by LOCF)
Population: FAS population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Synvisc
Number analyzed (Participants) | 232
mm
  Change form baseline at Week 8 | -26.0 (17.68)
  Change form baseline at Week 12 | -30.0 (17.43)

4. Secondary Outcome: Change From Baseline in WOMAC A, B and C Score at Weeks 8, 12 and 26
Description: WOMAC is health status measure questionnaire of twenty-four questions comprising 3 subscales (pain, stiffness and physical function). Each question was measured on a scale of 0-100 mm where lower score represents lower pain (better condition) and higher score represents higher pain. WOMAC A (measure of pain during walking on a flat surface) was sum of first five items with total score ranging from 0-500 mm, Lower score represents lower pain and higher score represents higher pain. WOMAC B (Stiffness) is the sum of the sixth and seventh item, it is in the range of 0-200 mm. WOMAC C (function) is the sum of the eighth to twenty-forth item, the score is in the range of 0-1700 mm.
Time Frame: Baseline, Week 8, 12 and 26 (missing data imputed by LOCF)
Population: FAS population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Synvisc
Number analyzed (Participants) | 232
mm
  WOMAC A: Change from baseline at Week 8 | -92.7 (71.77)
  WOMAC A: Change from baseline at Week 12 | -109.8 (73.68)
  WOMAC A: Change from baseline at Week 26 | -121.5 (77.18)
  WOMAC B: Change from baseline at Week 8 | -28.9 (37.53)
  WOMAC B: Change from baseline at Week 12 | -34.6 (38.44)
  WOMAC B: Change from baseline at Week 26 | -36.6 (39.75)
  WOMAC C: Change from baseline at Week 8 | -270.0 (252.86)
  WOMAC C: Change from baseline at Week 12 | -325.9 (258.57)
  WOMAC C: Change from baseline at Week 26 | -358.4 (270.48)

5. Secondary Outcome: Patient Global Assessment (PTGA) Score
Description: PTGA (self-assessment of target knee osteoarthritis condition) was measured using the 5 point Likert scale (0=very well, 1=well, 2=fair, 3=poor, 4=very poor) by participants to rate the osteoarthritis condition. Percentage of participants with different categories of PTGA score at baseline, Week 8, 12 and 26 are reported.
Time Frame: Baseline, Week 8, 12 and 26 (missing data imputed by LOCF)
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Synvisc
Number analyzed (Participants) | 232
percentage of participants
  Baseline: Very Well | 0.0
  Baseline: Well | 1.3
  Baseline: Fair | 29.3
  Baseline: Poor | 60.3
  Baseline: Very Poor | 9.1
  Week 8: Very Well | 4.3
  Week 8: Well | 41.8
  Week 8: Fair | 46.1
  Week 8 : Poor | 6.9
  Week 8: Very Poor | 0.9
  Week 12: Very Well | 5.2
  Week 12: Well | 44.4
  Week 12: Fair | 44.0
  Week 12: Poor | 6.0
  Week 12: Very Poor | 0.4
  Week 26: Very Well | 8.2
  Week 26: Well | 46.6
  Week 26: Fair | 37.1
  Week 26: Poor | 7.8
  Week 26: Very Poor | 0.4

6. Secondary Outcome: Clinical Observer Global Assessment (COGA) Score
Description: COGA (assessment of target knee osteoarthritis condition) was measured using the 5 point Likert scale (0=very well, 1=well, 2=fair, 3=poor, 4=very poor) by the physician to rate participant's osteoarthritis condition. Percentage of participants with different categories of COGA score at baseline,Week 8, 12 and 26 are reported.
Time Frame: Baseline, Week 8, 12 and 26 (missing data imputed by LOCF)
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Synvisc
Number analyzed (Participants) | 232
percentage of participants
  Baseline: Very Well | 0.0
  Baseline: Well | 1.7
  Baseline: Fair | 35.3
  Baseline: Poor | 57.3
  Baseline: Very Poor | 5.6
  Week 8: Very Well | 5.2
  Week 8: Well | 42.7
  Week 8: Fair | 41.8
  Week 8: Poor | 9.9
  Week 8: Very Poor | 0.4
  Week 12: Very Well | 7.3
  Week 12: Well | 44.4
  Week 12: Fair | 41.8
  Week 12: Poor | 6.0
  Week 12: Very Poor | 0.4
  Week 26: Very Well | 9.5
  Week 26: Well | 47.4
  Week 26: Fair | 35.3
  Week 26: Poor | 7.8
  Week 26: Very Poor | 0.0

7. Secondary Outcome: Percentage of Participants With Change in Concomitant Medication of Osteoarthritis Therapy at Week 26
Description: Participants were asked about their perception regarding any additional Osteoarthritis medications or treatments or any changes in regimen or dosages compared to their baseline (Day 1) state. Any change in the therapy (less use of other therapies, more use of other therapies and no change in use of other therapies) during the study was reported.
Time Frame: Baseline up to Week 26
Population: FAS population.
Measure: Number; unit: percentage participants
Arm/Group | Synvisc
Number analyzed (Participants) | 232
percentage participants
  Required Less Use of Other Therapies | 2.2
  Required More Use of Other Therapies | 3.0
  Required No Change in Use of Other Therapies | 93.1
  Missing | 1.7

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 26) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the time of signing the informed consent until completion of the study).
Arm/Group | Synvisc
Serious Adverse Events (participants affected / at risk) | 4/237
Other Adverse Events (participants affected / at risk) | 66/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc (N=237)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Meniscal Injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc (N=237)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Amyasthenia (Musculoskeletal and connective tissue disorders) | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1
Extremitiess Pain (Musculoskeletal and connective tissue disorders) | 1
Vertebral Disc Prolapsed (Musculoskeletal and connective tissue disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 17
Urinary Tract Infection (Infections and infestations) | 3
Herpes Zoster (Infections and infestations) | 1
Hand Infection (Infections and infestations) | 1
Infectious Pneumonia (Infections and infestations) | 1
Pain in the Area of Injection Site (General disorders) | 5
Weakness (General disorders) | 2
Swelling in the Area of Injection Site (General disorders) | 2
Warmth (General disorders) | 1
Joint Effusion in the Area of Injection Site (General disorders) | 1
Astriction (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Colonic Polyp (Gastrointestinal disorders) | 1
Atrophic Gastritis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Ligament Spain (Injury, poisoning and procedural complications) | 4
Meniscal Injury (Injury, poisoning and procedural complications) | 1
Extremities Injury (Injury, poisoning and procedural complications) | 1
Humeral Fracture (Injury, poisoning and procedural complications) | 1
Night Sweat (Skin and subcutaneous tissue disorders) | 1
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Migraine (Psychiatric disorders) | 1
Dizziness (Psychiatric disorders) | 1
Cramp (Psychiatric disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Colporrhagia (Reproductive system and breast disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Retinal Hemorrhage (Eye disorders) | 1
Gastritis (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.